CLINICAL TRIAL: NCT01995435
Title: Refraction Determination Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lee, Steven, M.D. (Individual)
Responsible Party: Principal Investigator, Coad Dow, MD, Investigator, Chippewa Valley Eye Clinic
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: SPL-321-REF
Record Dates: First submitted 2013-11-12; First posted 2013-11-26 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Myopia,; Hyperopia,; Astigmatism,; Presbyopia,; Eye Strain,
MeSH Terms: conditions — Myopia; Hyperopia; Astigmatism; Presbyopia; Asthenopia | interventions — Eyeglasses; Contact Lenses; Refractive Surgical Procedures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Telemedicine refraction before traditional refraction (Experimental): We will first refract an individual using telemedicine refraction, and then refract them using a traditional refraction method.
  Interventions: Device: Telemedicine refraction; Device: Traditional refraction
- Traditional refraction before telemedicine refraction (Experimental): We will first refract an individual using a traditional refraction, and then refract them using a telemedicine refraction method.
  Interventions: Device: Telemedicine refraction; Device: Traditional refraction

INTERVENTIONS:
Device: Telemedicine refraction
  Other Names: Glasses,; Contact lenses,; Refractive surgery,
Device: Traditional refraction

SUMMARY:
Correlating the accuracy of a refraction done over telemedicine to that of a standard refraction, with a study hypothesis that the results will be equivalent.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old
* healthy eyes

Exclusion Criteria:

* mid level ocular diseases (glaucoma, hypertension, retinal issues)
* psychiatric disorders
* brain tumor or history of
* under 18, or over 40 years old

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
refraction in diopters over telemedicine compared standard phoropter refraction | an average of 1 year

SECONDARY OUTCOMES:
telemedicine refraction results beyond dioptric readings | an average of 1 year
  to see if there are other uses for telemedicine refraction results

OTHER OUTCOMES:
patient satisfaction from telerefraction | an average of 1 year